CLINICAL TRIAL: NCT01097629
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of MK-4305 in Patients With Primary Insomnia - Study B
Brief Title: Safety and Efficacy Study of Suvorexant in Participants With Primary Insomnia - Study B (MK-4305-029)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4305-029; 2010_521 (Other: Merck Registration Number); CTRI/2010/091/001177 (Registry Identifier: CTRI)
Record Dates: First submitted 2010-03-26; First posted 2010-04-01 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Suvorexant HD (Experimental): Drug
  Interventions: Drug: Suvorexant High Dose (HD)
- Suvorexant LD (Experimental): Drug
  Interventions: Drug: Suvorexant Low Dose (LD)
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Suvorexant High Dose (HD) — Suvorexant 40 mg + placebo matching suvorexant 20 mg for participants <65 years old; Suvorexant 30 mg + placebo matching suvorexant 15 mg for participants ≥65 years old; all study drug is tablet for oral administration, taken once daily at bedtime. Participants receive this dose during the 3-month Treatment (TRT) Phase. During the 1-week double-blind (DB) Run-out (RO) following the TRT phase, participants in this study arm receive the noted suvorexant dose or placebo, in a 1:1 ratio. During the 2-week single-blind Run-in period prior to randomization all participants receive placebo to suvorexant once daily at bedtime.
  Other Names: MK-4305
  Arms: Suvorexant HD
Drug: Suvorexant Low Dose (LD) — Suvorexant 20 mg + placebo matching suvorexant 40 mg for participants <65 years old; Suvorexant 15 mg + placebo matching suvorexant 30 mg for participants ≥65 years old; all study drug is tablet for oral administration, taken once daily at bedtime. Participants receive this dose during the 3-month TRT Phase. During the 1-week DB RO following the TRT phase, participants in this study arm receive the noted suvorexant dose or placebo, in a 1:1 ratio. During the 2-week single-blind Run-in period prior to randomization all participants receive placebo to suvorexant once daily at bedtime.
  Other Names: MK-4305
  Arms: Suvorexant LD
Drug: Comparator: Placebo — Matching placebos to suvorexant 40 mg and 20 mg for participants <65 years old; matching placebos to suvorexant 30 mg and 15 mg for participants ≥65 years old; all study drug is tablet for oral administration, taken once daily at bedtime. Placebo is a third treatment arm for comparison to the two active (suvorexant) treatment arms during the 3-month TRT Phase. During the 1-week DB RO following the TRT phase, participants in this study arm continue to receive placebo. During the 2-week single-blind Run-in period prior to randomization all participants receive placebo to suvorexant once daily at bedtime.
  Arms: Placebo

SUMMARY:
This is a multicenter study to test the hypothesis that suvorexant (MK-4305) is superior to placebo in improving insomnia as measured by change from baseline in: subjective total sleep time and time to sleep onset, wake time after persistent sleep onset, and latency to onset of persistent sleep.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥18 yrs old on the day of signing informed consent
* Diagnosed with Primary Insomnia
* Good physical and mental health
* Participant ≥65 yrs old score at least 25 on the Mini Mental State Examination
* A female participant who is of reproductive potential has a negative serum pregnancy test and agrees to use contraception
* Reports difficulty with initiating and maintaining sleep during the 4 weeks prior to Visit 1 (accordingly to specific protocol criteria)
* Reports spending 6.5 to 9 hours nightly in bed on at least 3 out of 7 nights prior to Visit 1
* Regular bedtime is between 9 pm-1 am
* Willing to refrain from napping while in study
* Able to read, understand and complete questionnaires and all diaries
* Willing to limit alcohol, caffeine, and nicotine consumption while in the study
* For a portion of participants: Must be willing to stay overnight in a sleep laboratory and must be willing to stay in bed for at least 8 hours each night while at the sleep laboratory

Exclusion Criteria:

* Female participant is pregnant and/or breastfeeding at Prestudy visit, or expecting to conceive while in study
* History or diagnosis of another sleep disorder
* Difficulty sleeping due to a medical condition
* History of a neurological disorder
* History of bipolar disorder, psychotic disorder, or posttraumatic stress disorder, or current psychiatric disorder that requires a prohibited medication
* Ongoing depression
* History of substance abuse or dependence
* History or current evidence of a clinically significant cardiovascular disorder or clinically significant electrocardiogram (ECG) at Prestudy Visit
* Taking certain prohibited medications
* Consumption of the equivalent of >15 cigarettes a day
* History of malignancy ≤5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* Participant is considered morbidly obese
* Previously randomized in another investigational study of suvorexant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Actual)
Dates: Start 2010-05-03 (Actual); Primary Completion 2011-11-08 (Actual); Study Completion 2011-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Herring WJ, Connor KM, Ivgy-May N, Snyder E, Liu K, Snavely DB, Krystal AD, Walsh JK, Benca RM, Rosenberg R, Sangal RB, Budd K, Hutzelmann J, Leibensperger H, Froman S, Lines C, Roth T, Michelson D. Suvorexant in Patients With Insomnia: Results From Two 3-Month Randomized Controlled Clinical Trials. Biol Psychiatry. 2016 Jan 15;79(2):136-48. doi: 10.1016/j.biopsych.2014.10.003. Epub 2014 Oct 23. PMID 25526970
- [Derived] Tao P, Svetnik V, Bliwise DL, Zammit G, Lines C, Herring WJ. Comparison of polysomnography in people with Alzheimer's disease and insomnia versus non-demented elderly people with insomnia. Sleep Med. 2023 Jan;101:515-521. doi: 10.1016/j.sleep.2022.11.027. Epub 2022 Dec 1. PMID 36529106
- [Derived] Snyder ES, Tao P, Svetnik V, Lines C, Herring WJ. Use of the single-item Patient Global Impression-Severity scale as a self-reported assessment of insomnia severity. J Sleep Res. 2021 Feb;30(1):e13141. doi: 10.1111/jsr.13141. Epub 2020 Jul 30. PMID 33210445
- [Derived] Svetnik V, Snyder ES, Tao P, Roth T, Lines C, Herring WJ. How well can a large number of polysomnography sleep measures predict subjective sleep quality in insomnia patients? Sleep Med. 2020 Mar;67:137-146. doi: 10.1016/j.sleep.2019.08.020. Epub 2019 Sep 11. PMID 31926466
- [Derived] Herring WJ, Connor KM, Snyder E, Snavely DB, Morin CM, Lines C, Michelson D. Effects of suvorexant on the Insomnia Severity Index in patients with insomnia: analysis of pooled phase 3 data. Sleep Med. 2019 Apr;56:219-223. doi: 10.1016/j.sleep.2018.09.010. Epub 2018 Oct 2. PMID 30522875
- [Derived] Svetnik V, Snyder ES, Tao P, Scammell TE, Roth T, Lines C, Herring WJ. Insight Into Reduction of Wakefulness by Suvorexant in Patients With Insomnia: Analysis of Wake Bouts. Sleep. 2018 Jan 1;41(1). doi: 10.1093/sleep/zsx178. PMID 29112763
- [Derived] Herring WJ, Connor KM, Snyder E, Snavely DB, Zhang Y, Hutzelmann J, Matzura-Wolfe D, Benca RM, Krystal AD, Walsh JK, Lines C, Roth T, Michelson D. Suvorexant in Elderly Patients with Insomnia: Pooled Analyses of Data from Phase III Randomized Controlled Clinical Trials. Am J Geriatr Psychiatry. 2017 Jul;25(7):791-802. doi: 10.1016/j.jagp.2017.03.004. Epub 2017 Mar 8. PMID 28427826
- [Derived] Herring WJ, Connor KM, Snyder E, Snavely DB, Zhang Y, Hutzelmann J, Matzura-Wolfe D, Benca RM, Krystal AD, Walsh JK, Lines C, Roth T, Michelson D. Clinical profile of suvorexant for the treatment of insomnia over 3 months in women and men: subgroup analysis of pooled phase-3 data. Psychopharmacology (Berl). 2017 Jun;234(11):1703-1711. doi: 10.1007/s00213-017-4573-1. Epub 2017 Mar 7. PMID 28265715
- [Derived] Herring WJ, Connor KM, Snyder E, Snavely DB, Zhang Y, Hutzelmann J, Matzura-Wolfe D, Benca RM, Krystal AD, Walsh JK, Lines C, Roth T, Michelson D. Suvorexant in Patients with Insomnia: Pooled Analyses of Three-Month Data from Phase-3 Randomized Controlled Clinical Trials. J Clin Sleep Med. 2016 Sep 15;12(9):1215-25. doi: 10.5664/jcsm.6116. PMID 27397664
- [Derived] Snyder E, Ma J, Svetnik V, Connor KM, Lines C, Michelson D, Herring WJ. Effects of suvorexant on sleep architecture and power spectral profile in patients with insomnia: analysis of pooled phase 3 data. Sleep Med. 2016 Mar;19:93-100. doi: 10.1016/j.sleep.2015.10.007. Epub 2015 Nov 10. PMID 27198953
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=4305-029&kw=4305-029&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A 2-week single-blind placebo Run-in occurred prior to randomization. 1 of the 1020 randomized participants enrolled in 2 separate suvorexant trials and is excluded from all summaries and analyses. 10 other randomized participants were not treated and are in Participant Flow Table below, but are excluded from all other summaries and analyses.
Groups:
- Suvorexant Low Dose (LD) (TRT Phase): After a 2-week single-blind placebo Run-in, participants received suvorexant LD (20 mg for participants aged 18 to <65 years; and 15 mg for participants aged ≥65 years) daily before bedtime during the 3-month DB TRT Phase.
- Suvorexant High Dose (HD) (TRT Phase): After a 2-week single-blind placebo Run-in, participants received suvorexant HD (40 mg for participants aged 18 to <65 years; and 30 mg for participants aged ≥65 years) daily before bedtime during the 3-month DB TRT Phase.
- Placebo (TRT Phase): After a 2-week single-blind placebo Run-in, participants received placebo to suvorexant daily before bedtime during the 3-month double-blind DB TRT Phase.
- Suvorexant LD (Run-out [RO], After Suvorexant LD in TRT): After receiving suvorexant LD during the 3-Month DB TRT Phase, participants received their same dose of suvorexant during a 1-week DB RO Phase.
- Placebo (RO, After Suvorexant LD in TRT): After receiving suvorexant LD during the 3-Month DB TRT Phase, participants received placebo to suvorexant during a 1-week DB RO Phase.
- Suvorexant HD (RO, After Suvorexant HD in TRT): After receiving suvorexant HD during the 3-Month DB TRT Phase, participants received their same dose of suvorexant during a 1-week DB RO Phase.
- Placebo (RO, After Suvorexant HD in TRT): After receiving suvorexant HD during the 3-Month DB TRT Phase, participants received placebo to suvorexant during a 1-week DB RO Phase.
- Placebo (RO, After Placebo in TRT): After receiving placebo to suvorexant during the 3-Month DB TRT Phase, participants received placebo to suvorexant during a 1-week DB RO Phase.
Period: Double-Blind (DB) Treatment (TRT) Phase
Arm/Group | Suvorexant Low Dose (LD) (TRT Phase) | Suvorexant High Dose (HD) (TRT Phase) | Placebo (TRT Phase) | Suvorexant LD (Run-out [RO], After Suvorexant LD in TRT) | Placebo (RO, After Suvorexant LD in TRT) | Suvorexant HD (RO, After Suvorexant HD in TRT) | Placebo (RO, After Suvorexant HD in TRT) | Placebo (RO, After Placebo in TRT)
Started | 240 | 392 | 387 | 0 | 0 | 0 | 0 | 0
Treated | 239 | 387 | 383 | 0 | 0 | 0 | 0 | 0
Completed | 205 | 346 (2 did not continue into RO) | 330 (3 did not continue into RO) | 0 | 0 | 0 | 0 | 0
Not Completed | 35 | 46 | 57 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 19 | 17 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 9 | 19 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 5 | 4 | 8 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 7 | 4 | 8 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not Treated | 1 | 5 | 4 | 0 | 0 | 0 | 0 | 0
Period: DB RO Phase
Arm/Group | Suvorexant Low Dose (LD) (TRT Phase) | Suvorexant High Dose (HD) (TRT Phase) | Placebo (TRT Phase) | Suvorexant LD (Run-out [RO], After Suvorexant LD in TRT) | Placebo (RO, After Suvorexant LD in TRT) | Suvorexant HD (RO, After Suvorexant HD in TRT) | Placebo (RO, After Suvorexant HD in TRT) | Placebo (RO, After Placebo in TRT)
Started | 0 | 0 | 0 | 97 | 108 | 173 | 171 | 327
Completed | 0 | 0 | 0 | 96 | 108 | 172 | 168 | 326
Not Completed | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Suvorexant LD: After a 2-week single-blind placebo Run-in, participants received suvorexant LD (20 mg for participants aged 18 to <65 years; and 15 mg for participants aged ≥65 years) daily before bedtime during the 3-month DB TRT Phase.
- Suvorexant HD: After a 2-week single-blind placebo Run-in, participants received suvorexant HD (40 mg for participants aged 18 to <65 years; and 30 mg for participants aged ≥65 years) daily before bedtime during the 3-month DB TRT Phase.
- Placebo: After a 2-week single-blind placebo Run-in, participants received placebo to suvorexant daily before bedtime during the 3-month double-blind DB TRT Phase.
- Total: Total of all reporting groups
Arm/Group | Suvorexant LD | Suvorexant HD | Placebo | Total
Number analyzed (Participants) | 239 | 387 | 383 | 1009
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (16) | 57 (15) | 57 (15) | 56 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 267 | 247 | 671
  Male | 82 | 120 | 136 | 338
Mean Subjective Total Sleep Time (sTSTm) [Mean (Standard Deviation); unit: minutes] — N=238, 386, 383, 1007 for Suvorexant Low Dose, Suvorexant High Dose, Placebo and Total, respectively.
  minutes | 298.3 (81.9) | 315.3 (77.0) | 309.7 (77.1) | 309.2 (78.4)
Wakefulness After Persistent Sleep Onset (WASO) [Mean (Standard Deviation); unit: minutes] — N=150, 299, 295, 744 for Suvorexant Low Dose, Suvorexant High Dose, Placebo and Total, respectively. WASO was assessed during sleep laboratory (polysomnography [PSG]) assessment, which was conducted in a subset of the study population.
  minutes | 119.6 (50.8) | 119.4 (51.3) | 118.4 (49.1) | 119.0 (50.3)
Mean Subjective Time to Sleep Onset (sTSOm) [Mean (Standard Deviation); unit: minutes] — N=238, 386, 383, 1007 for Suvorexant Low Dose, Suvorexant High Dose, Placebo and Total, respectively.
  minutes | 86.0 (77.6) | 74.4 (61.9) | 81.3 (76.2) | 79.8 (71.5)
Latency to Onset of Persistent Sleep (LPS) [Mean (Standard Deviation); unit: minutes] — N=150, 299, 295, 744 for Suvorexant Low Dose, Suvorexant High Dose, Placebo and Total, respectively. LPS was assessed during sleep laboratory (PSG) assessment, which was conducted in a subset of the study population.
  minutes | 65.3 (47.8) | 67.3 (48.8) | 68.0 (42.8) | 67.2 (46.2)

OUTCOME MEASURES:

1. Primary Outcome: Suvorexant HD Versus Placebo: Change From Baseline in Mean Subjective Total Sleep Time (sTSTm) at Month 1
Description: sTSTm is the average over a defined day range of the participant's report of the total amount of time spent asleep before waking for the day, as recorded in a daily electronic diary (e-diary). Averages were derived by taking the mean of all available daily measurements (excluding the mornings following any polysomnography [PSG] nights) falling within the day range; Month 1 range is Days 23-30 (Day 1 is day of first double-blind dose). A participant must have at least 3 days of data during the defined day range to calculate an average for the day range; otherwise, the mean value was considered missing for that day range. The baseline value is the mean of the last 7 daily measurements obtained during the placebo Run-in period.
Time Frame: Baseline and Month 1
Population: Randomized participants with ≥1 post-randomization e-diary observation after ≥1 dose of study drug, and baseline data were included in this analysis. The hypothesis included only the suvorexant HD-placebo comparison.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant HD | Placebo
Number analyzed (Participants) | 365 | 350
minutes | 48.7 (77.4) [43.1 to 54.3] | 22.4 (77.6) [16.7 to 28.1]
Statistical Analysis 1: Comparison: Suvorexant HD vs Placebo; The null hypothesis, that suvorexant HD did not differ from placebo for Month 1 sTSTm, had planned marginal power of 97.6%. Sleep maintenance (sTSTm, WASO) and sleep onset (sTSOm, LPS) endpoints were tested at two-sided 2.5% significance level. Both Month 1 endpoints for sleep maintenance must be significant to test Month 3 endpoints; the same approach was used for sleep onset endpoints; Test type: Superiority or Other; p < 0.00001, Longitudinal Data Analysis — By multiplicity strategy above, overall Type I error among primary hypotheses was controlled at two-sided 5% significance level; Model terms: baseline value, age group, region, gender, treatment, time, time by treatment interaction, and cohort (e-diary only, PSG-plus-e-diary); Difference in Least Squares Means = 26.3, 95% CI 2-sided [18.3 to 34.3]

2. Primary Outcome: Suvorexant HD Versus Placebo: Change From Baseline in sTSTm at Month 3
Description: sTSTm is the average over a defined day range of the participant's report of the total amount of time spent asleep before waking for the day, as recorded in a daily e-diary. Averages were derived by taking the mean of all available daily measurements (excluding the mornings following any PSG nights) falling within the day range; Month 3 range is Days 76-90 (Day 1 is day of first double-blind dose). A participant must have at least 3 days of data during the defined day range to calculate an average for the day range; otherwise, the mean value was considered missing for that day range. The baseline value is the mean of the last 7 daily measurements obtained during the placebo Run-in period.
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant HD | Placebo
Number analyzed (Participants) | 340 | 325
minutes | 62.8 (75.9) [56.4 to 69.2] | 37.7 (71.8) [31.2 to 44.2]
Statistical Analysis 1: Comparison: Suvorexant HD vs Placebo; The null hypothesis, that suvorexant HD did not differ from placebo for Month 3 sTSTm, had planned marginal power of 95.7%. Sleep maintenance (sTSTm, WASO) and sleep onset (sTSOm, LPS) endpoints were tested at two-sided 2.5% significance level. Both Month 1 endpoints for sleep maintenance must be significant to test Month 3 endpoints; the same approach was used for sleep onset endpoints; Test type: Superiority or Other; p < 0.00001, Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 25.1, 95% CI [16.0 to 34.2]

3. Primary Outcome: Suvorexant HD Versus Placebo: Change From Baseline in Wakefulness After Persistent Sleep Onset (WASO) at Month 1
Description: WASO is measured during overnight sleep laboratory (PSG) assessments at baseline, Night 1, Month 1 and Month 3, and is defined as the duration of wakefulness from the onset of persistent sleep (i.e., 10 consecutive minutes of sleep) to the end of PSG assessment the following morning. Beginning of PSG assessment ("Lights-Off") is at approximately the participant's habitual bedtime. The participant is awakened, or allowed to get out of bed if already awake, after 8 hours of PSG recording ("Lights-On"). PSG assessments consist of electronic measurement of brain activity and eye and muscle movements. PSG data was scored by a Centralized PSG reading center.
Time Frame: Baseline and Month 1
Population: Randomized participants with ≥1 post-randomization PSG observation after ≥1 dose of study drug, and baseline data were included in this analysis. The hypothesis included only the suvorexant HD-placebo comparison.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant HD | Placebo
Number analyzed (Participants) | 278 | 270
minutes | -51.9 (51.2) [-56.9 to -46.9] | -22.5 (49.3) [-27.5 to -17.4]
Statistical Analysis 1: Comparison: Suvorexant HD vs Placebo; The null hypothesis, that suvorexant HD did not differ from placebo for Month 1 WASO, had planned marginal power of 99.2%. Sleep maintenance (sTSTm, WASO) and sleep onset (sTSOm, LPS) endpoints were tested at two-sided 2.5% significance level. Both Month 1 endpoints for sleep maintenance must be significant to test Month 3 endpoints; the same approach was used for sleep onset endpoints; Test type: Superiority or Other; p < 0.00001, Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Model terms: baseline value, age group, region, gender, treatment, time, and time by treatment interaction; Difference in Least Squares Means = -29.4, 95% CI 2-sided [-36.6 to -22.3]

4. Primary Outcome: Suvorexant HD Versus Placebo: Change From Baseline in WASO at Month 3
Description: as for outcome 3
Time Frame: Baseline and Month 3
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant HD | Placebo
Number analyzed (Participants) | 260 | 252
minutes | -54.2 (51.1) [-59.3 to -49.1] | -24.8 (49.6) [-30.0 to -19.6]
Statistical Analysis 1: Comparison: Suvorexant HD vs Placebo; The null hypothesis, that suvorexant HD did not differ from placebo for Month 3 WASO, had planned marginal power of 98.3%. Sleep maintenance (sTSTm, WASO) and sleep onset (sTSOm, LPS) endpoints were tested at two-sided 2.5% significance level. Both Month 1 endpoints for sleep maintenance must be significant to test Month 3 endpoints; the same approach was used for sleep onset endpoints; Test type: Superiority or Other; p < 0.00001, Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Model terms: baseline value, age group, region, gender, treatment, time, and time by treatment interaction; Difference in Least Squares Means = -29.4, 95% CI 2-sided [-36.7 to -22.1]

5. Primary Outcome: Suvorexant HD Versus Placebo: Change From Baseline in Mean Subjective Time to Sleep Onset (sTSOm) at Month 1
Description: sTSOm is the average over a defined day range of the participant's report of the duration of time that it took to fall asleep, as recorded in a daily e-diary. Averages were derived by taking the mean of all available daily measurements (excluding the mornings following any PSG nights) falling within the day range; Month 1 range is Days 23-30 (Day 1 is day of first double-blind dose). A participant must have at least 3 days of data during the defined day range to calculate an average for the day range; otherwise, the mean value was considered missing for that day range. The baseline value is the mean of the last 7 daily measurements obtained during the placebo Run-in period.
Time Frame: Baseline and Month 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant HD | Placebo
Number analyzed (Participants) | 365 | 350
minutes | -26.9 (62.8) [-31.1 to -22.8] | -14.1 (77.8) [-18.4 to -9.9]
Statistical Analysis 1: Comparison: Suvorexant HD vs Placebo; The null hypothesis, that suvorexant HD did not differ from placebo for Month 1 sTSOm, had planned marginal power of 99.9%. Sleep maintenance (sTSTm, WASO) and sleep onset (sTSOm, LPS) endpoints were tested at two-sided 2.5% significance level. Both Month 1 endpoints for sleep maintenance must be significant to test Month 3 endpoints; the same approach was used for sleep onset endpoints; Test type: Superiority or Other; p = 0.00003, Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -12.8, 95% CI 2-sided [-18.8 to -6.9]

6. Primary Outcome: Suvorexant HD Versus Placebo: Change From Baseline in sTSOm at Month 3
Description: sTSOm is the average over a defined day range of the participant's report of the duration of time that it took to fall asleep, as recorded in a daily e-diary. Averages were derived by taking the mean of all available daily measurements (excluding the mornings following any PSG nights) falling within the day range; Month 3 range is Days 76-90 (Day 1 is day of first double-blind dose). A participant must have at least 3 days of data during the defined day range to calculate an average for the day range; otherwise, the mean value was considered missing for that day range. The baseline value is the mean of the last 7 daily measurements obtained during the placebo Run-in period.
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant HD | Placebo
Number analyzed (Participants) | 340 | 325
minutes | -33.7 (62.4) [-38.0 to -29.3] | -20.5 (66.1) [-24.9 to -16.1]
Statistical Analysis 1: Comparison: Suvorexant HD vs Placebo; The null hypothesis, that suvorexant HD did not differ from placebo for Month 3 sTSOm, had planned marginal power of 99.6%. Sleep maintenance (sTSTm, WASO) and sleep onset (sTSOm, LPS) endpoints were tested at two-sided 2.5% significance level. Both Month 1 endpoints for sleep maintenance must be significant to test Month 3 endpoints; the same approach was used for sleep onset endpoints; Test type: Superiority or Other; p = 0.00003, Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -13.2, 95% CI 2-sided [-19.4 to -7.0]

7. Primary Outcome: Suvorexant HD Versus Placebo: Change From Baseline in Latency to Onset of Persistent Sleep (LPS) at Month 1
Description: LPS is measured during overnight sleep laboratory (PSG) assessments at baseline, Night 1, Month 1 and Month 3, and is defined as the duration of time from the beginning of PSG assessment ("Lights-Off") to the first interval of 10 consecutive minutes of sleep. Beginning of PSG assessment ("Lights-Off") is at approximately the participant's habitual bedtime. The participant is awakened, or allowed to get out of bed if already awake, after 8 hours of PSG recording ("Lights-On"). PSG assessments consist of electronic measurement of brain activity and eye and muscle movements. PSG data was scored by a Centralized PSG reading center.
Time Frame: Baseline and Month 1
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant HD | Placebo
Number analyzed (Participants) | 280 | 271
minutes | -36.7 (46.5) [-40.8 to -32.7] | -24.6 (43.3) [-28.7 to -20.6]
Statistical Analysis 1: Comparison: Suvorexant HD vs Placebo; The null hypothesis, that suvorexant HD did not differ from placebo for Month 1 LPS, had planned marginal power of 81.4%. Sleep maintenance (sTSTm, WASO) and sleep onset (sTSOm, LPS) endpoints were tested at two-sided 2.5% significance level. Both Month 1 endpoints for sleep maintenance must be significant to test Month 3 endpoints; the same approach was used for sleep onset endpoints; Test type: Superiority or Other; p = 0.00004, Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Model terms: baseline value, age group, region, gender, treatment, time, and time by treatment interaction; Difference in Least Squares Means = -12.1, 95% CI 2-sided [-17.8 to -6.4]

8. Primary Outcome: Suvorexant HD Versus Placebo: Change From Baseline in LPS at Month 3
Description: as for outcome 7
Time Frame: Baseline and Month 3
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant HD | Placebo
Number analyzed (Participants) | 262 | 255
minutes | -32.2 (47.6) [-36.7 to -27.7] | -28.6 (44.0) [-33.1 to -24.0]
Statistical Analysis 1: Comparison: Suvorexant HD vs Placebo; The null hypothesis, that suvorexant HD did not differ from placebo for Month 3 LPS, had planned marginal power of 76.2%. Sleep maintenance (sTSTm, WASO) and sleep onset (sTSOm, LPS) endpoints were tested at two-sided 2.5% significance level. Both Month 1 endpoints for sleep maintenance must be significant to test Month 3 endpoints; the same approach was used for sleep onset endpoints; Test type: Superiority or Other; p = 0.26510, Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Model terms: baseline value, age group, region, gender, treatment, time, and time by treatment interaction; Difference in Least Squares Means = -3.6, 95% CI 2-sided [-10.1 to 2.8]

9. Secondary Outcome: Suvorexant HD Versus Placebo: Change From Baseline in sTSTm at Week 1
Description: sTSTm is the average over a defined day range of the participant's report of the total amount of time spent asleep before waking for the day, as recorded in a daily e-diary. Averages were derived by taking the mean of all available daily measurements (excluding the mornings following any PSG nights) falling within the day range; Week 1 range is Days 2-8 (Day 1 is day of first double-blind dose). A participant must have at least 3 days of data during the defined day range to calculate an average for the day range; otherwise, the mean value was considered missing for that day range. The baseline value is the mean of the last 7 daily measurements obtained during the placebo Run-in period.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant HD | Placebo
Number analyzed (Participants) | 373 | 364
minutes | 40.4 (83.1) [35.7 to 45.1] | 14.0 (81.0) [9.2 to 18.7]
Statistical Analysis 1: Comparison: Suvorexant HD vs Placebo; The null hypothesis, that suvorexant HD did not differ from placebo for Week 1 sTSTm, had planned marginal power of 98.3%. Sleep maintenance (sTSTm, WASO) and sleep onset (sTSOm, LPS) endpoints were tested at two-sided 2.5% significance level. Both Month 1 endpoints for sleep maintenance must be significant to test Month 3 endpoints and either subjective or objective Month 3 endpoint must be significant to test Week 1/Night 1 endpoints. The same approach was used for sleep onset endpoints; Test type: Superiority or Other; p < 0.00001, Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 26.4, 95% CI 2-sided [19.8 to 33.1]

10. Secondary Outcome: Suvorexant HD Versus Placebo: Change From Baseline in WASO at Night 1
Description: as for outcome 3
Time Frame: Baseline and Night 1
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant HD | Placebo
Number analyzed (Participants) | 285 | 283
minutes | -63.3 (37.5) [-68.0 to -58.6] | -21.3 (65.5) [-26.1 to -16.6]
Statistical Analysis 1: Comparison: Suvorexant HD vs Placebo; The null hypothesis, that suvorexant HD did not differ from placebo for Night 1 WASO, had planned marginal power of 100.0%. Sleep maintenance (sTSTm, WASO) and sleep onset (sTSOm, LPS) endpoints were tested at two-sided 2.5% significance level. Both Month 1 endpoints for sleep maintenance must be significant to test Month 3 endpoints and either subjective or objective Month 3 endpoint must be significant to test Week 1/Night 1 endpoints. The same approach was used for sleep onset endpoints; Test type: Superiority or Other; p < 0.00001, Longitudinal Data Analysis; Model terms: baseline value, age group, region, gender, treatment, time, and time by treatment interaction; Difference in Least Squares Means = -42.0, 95% CI 2-sided [-48.6 to -35.3]

11. Secondary Outcome: Suvorexant HD Versus Placebo: Change From Baseline in sTSOm at Week 1
Description: sTSOm is the average over a defined day range of the participant's report of the duration of time that it took to fall asleep, as recorded in a daily e-diary. Averages were derived by taking the mean of all available daily measurements (excluding the mornings following any PSG nights) falling within the day range; Week 1 range is Days 2-8 (Day 1 is day of first double-blind dose). A participant must have at least 3 days of data during the defined day range to calculate an average for the day range; otherwise, the mean value was considered missing for that day range. The baseline value is the mean of the last 7 daily measurements obtained during the placebo Run-in period.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant HD | Placebo
Number analyzed (Participants) | 373 | 364
minutes | -19.7 (59.0) [-23.0 to -16.4] | -6.7 (76.0) [-10.0 to -3.3]
Statistical Analysis 1: Comparison: Suvorexant HD vs Placebo; The null hypothesis, that suvorexant HD did not differ from placebo for Week 1 sTSOm, had planned marginal power of 99.6%. Sleep maintenance (sTSTm, WASO) and sleep onset (sTSOm, LPS) endpoints were tested at two-sided 2.5% significance level. Both Month 1 endpoints for sleep maintenance must be significant to test Month 3 endpoints and either subjective or objective Month 3 endpoint must be significant to test Week 1/Night 1 endpoints. The same approach was used for sleep onset endpoints; Test type: Superiority or Other; p < 0.00001, Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -13.1, 95% CI 2-sided [-17.7 to -8.4]

12. Secondary Outcome: Suvorexant HD Versus Placebo: Change From Baseline in LPS at Night 1
Description: as for outcome 7
Time Frame: Baseline and Night 1
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant HD | Placebo
Number analyzed (Participants) | 289 | 284
minutes | -34.7 (24.2) [-39.5 to -29.9] | -13.0 (60.8) [-17.8 to -8.1]
Statistical Analysis 1: Comparison: Suvorexant HD vs Placebo; The null hypothesis, that suvorexant HD did not differ from placebo for Night 1 LPS, had planned marginal power of 100.0%. Sleep maintenance (sTSTm, WASO) and sleep onset (sTSOm, LPS) endpoints were tested at two-sided 2.5% significance level. Both Month 1 endpoints for sleep maintenance must be significant to test Month 3 endpoints and either subjective or objective Month 3 endpoint must be significant to test Week 1/Night 1 endpoints. The same approach was used for sleep onset endpoints; Test type: Superiority or Other; p < 0.00001, Longitudinal Data Analysis; Model terms: baseline value, age group, region, gender, treatment, time, and time by treatment interaction; Difference in Least Squares Means = -21.7, 95% CI 2-sided [-28.6 to -14.9]

13. Primary Outcome: Number of Participants With an Adverse Event (AE) During 3-Month DB TRT Phase
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug. Participants with an AE occurring during the 3-month DB TRT Phase are counted once in this summary.
Time Frame: Up to 3 months
Population: All Patients as Treated (APaT) population, consisting of all randomized participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Suvorexant LD | Suvorexant HD | Placebo
Number analyzed (Participants) | 239 | 387 | 383
participants | 103 | 189 | 167

14. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE Occurring During 3-Month DB TRT Phase
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug. Participants who discontinued study drug treatment due to an AE occurring during the 3-month DB TRT Phase are counted once in this summary.
Time Frame: Up to 3 months
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Suvorexant LD | Suvorexant HD | Placebo
Number analyzed (Participants) | 239 | 387 | 383
participants | 9 | 18 | 17

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last dose of study drug
Description: The 3 TRT Phase reporting groups include total population; other groups present same or subsets of this population in other study phases. Events are reported by phase. Phases are: - TRT - RO - Follow-up (enter directly from TRT Phase, or from RO)
Groups:
- Suvorexant LD (TRT Phase): After a 2-week single-blind placebo Run-in, participants received suvorexant LD (20 mg for participants aged 18 to <65 years; and 15 mg for participants aged ≥65 years) daily before bedtime during the 3-month DB TRT Phase.
- Suvorexant HD (TRT Phase): After a 2-week single-blind placebo Run-in, participants received suvorexant HD (40 mg for participants aged 18 to <65 years; and 30 mg for participants aged ≥65 years) daily before bedtime during the 3-month DB TRT Phase.
- Suvorexant LD (RO, After Suvorexant LD in TRT): After receiving suvorexant LD during the 3-Month DB TRT Phase, participants received their same dose of suvorexant during a 1-week DB RO Phase.
- Suvorexant LD (TRT Phase): Follow-up: During 14-day Follow-up after last dose no study drug was administered. Follow-up AE data is presented for TRT Phase participants who entered Follow-up directly from TRT Phase and had received suvorexant LD during TRT Phase.
- Suvorexant HD (TRT Phase): Follow-up: During 14-day Follow-up after last dose no study drug was administered. Follow-up AE data is presented for TRT Phase participants who entered Follow-up directly from TRT Phase and had received suvorexant HD during TRT Phase.
- Placebo (TRT Phase): Follow-up: During 14-day Follow-up after last dose no study drug was administered. Follow-up AE data is presented for TRT Phase participants who entered Follow-up directly from TRT Phase and had received placebo during TRT Phase.
- Suvorexant LD (RO, After Suvorexant LD in TRT): Follow-up: During 14-day Follow-up after last dose no study drug was administered. Follow-up AE data is presented for RO participants who entered Follow-up from RO Phase, and had received suvorexant LD during TRT and RO Phases.
- Placebo (RO, After Suvorexant LD in TRT): Follow-up: During 14-day Follow-up after last dose no study drug was administered. Follow-up AE data is presented for RO participants who entered Follow-up from RO Phase, and had received suvorexant LD during TRT Phase and placebo during RO Phase.
- Suvorexant HD (RO, After Suvorexant HD in TRT): Follow-up: During 14-day Follow-up after last dose no study drug was administered. Follow-up AE data is presented for RO participants who entered Follow-up from RO Phase, and had received suvorexant HD during TRT and RO Phases.
- Placebo (RO, After Suvorexant HD in TRT): Follow-up: During 14-day Follow-up after last dose no study drug was administered. Follow-up AE data is presented for RO participants who entered Follow-up from RO Phase, and had received suvorexant HD during TRT Phase and placebo during RO Phase.
- Placebo (RO, After Placebo in TRT): Follow-up: During 14-day Follow-up after last dose no study drug was administered. Follow-up AE data is presented for RO participants who entered Follow-up from RO Phase, and had received placebo during TRT and RO Phases.
Arm/Group | Suvorexant LD (TRT Phase) | Suvorexant HD (TRT Phase) | Placebo (TRT Phase) | Suvorexant LD (RO, After Suvorexant LD in TRT) | Placebo (RO, After Suvorexant LD in TRT) | Suvorexant HD (RO, After Suvorexant HD in TRT) | Placebo (RO, After Suvorexant HD in TRT) | Placebo (RO, After Placebo in TRT) | Suvorexant LD (TRT Phase): Follow-up | Suvorexant HD (TRT Phase): Follow-up | Placebo (TRT Phase): Follow-up | Suvorexant LD (RO, After Suvorexant LD in TRT): Follow-up | Placebo (RO, After Suvorexant LD in TRT): Follow-up | Suvorexant HD (RO, After Suvorexant HD in TRT): Follow-up | Placebo (RO, After Suvorexant HD in TRT): Follow-up | Placebo (RO, After Placebo in TRT): Follow-up
Serious Adverse Events (participants affected / at risk) | 2/239 | 6/387 | 5/383 | 0/97 | 1/108 | 0/173 | 0/171 | 0/327 | 0/239 | 1/387 | 0/383 | 0/97 | 0/108 | 0/173 | 0/171 | 0/327
Other Adverse Events (participants affected / at risk) | 33/239 | 59/387 | 33/383 | 0/97 | 1/108 | 4/173 | 1/171 | 4/327 | 0/239 | 2/387 | 0/383 | 0/97 | 1/108 | 0/173 | 0/171 | 1/327
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suvorexant LD (TRT Phase) (N=239) | Suvorexant HD (TRT Phase) (N=387) | Placebo (TRT Phase) (N=383) | Suvorexant LD (RO, After Suvorexant LD in TRT) (N=97) | Placebo (RO, After Suvorexant LD in TRT) (N=108) | Suvorexant HD (RO, After Suvorexant HD in TRT) (N=173) | Placebo (RO, After Suvorexant HD in TRT) (N=171) | Placebo (RO, After Placebo in TRT) (N=327) | Suvorexant LD (TRT Phase): Follow-up (N=239) | Suvorexant HD (TRT Phase): Follow-up (N=387) | Placebo (TRT Phase): Follow-up (N=383) | Suvorexant LD (RO, After Suvorexant LD in TRT): Follow-up (N=97) | Placebo (RO, After Suvorexant LD in TRT): Follow-up (N=108) | Suvorexant HD (RO, After Suvorexant HD in TRT): Follow-up (N=173) | Placebo (RO, After Suvorexant HD in TRT): Follow-up (N=171) | Placebo (RO, After Placebo in TRT): Follow-up (N=327)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
endometritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suvorexant LD (TRT Phase) (N=239) | Suvorexant HD (TRT Phase) (N=387) | Placebo (TRT Phase) (N=383) | Suvorexant LD (RO, After Suvorexant LD in TRT) (N=97) | Placebo (RO, After Suvorexant LD in TRT) (N=108) | Suvorexant HD (RO, After Suvorexant HD in TRT) (N=173) | Placebo (RO, After Suvorexant HD in TRT) (N=171) | Placebo (RO, After Placebo in TRT) (N=327) | Suvorexant LD (TRT Phase): Follow-up (N=239) | Suvorexant HD (TRT Phase): Follow-up (N=387) | Placebo (TRT Phase): Follow-up (N=383) | Suvorexant LD (RO, After Suvorexant LD in TRT): Follow-up (N=97) | Placebo (RO, After Suvorexant LD in TRT): Follow-up (N=108) | Suvorexant HD (RO, After Suvorexant HD in TRT): Follow-up (N=173) | Placebo (RO, After Suvorexant HD in TRT): Follow-up (N=171) | Placebo (RO, After Placebo in TRT): Follow-up (N=327)
headache (Nervous system disorders) | 19 (22) | 29 (32) | 22 (22) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
somnolence (Nervous system disorders) | 20 (21) | 40 (44) | 12 (13) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish results for his/her study site after publication of results of entire multicenter trial, or after public disclosure of the results online if a multicenter manuscript is not planned. Sponsor must be able to review all proposed results communications regarding study 60 days prior to submission for publication/presentation. Information identified by the Sponsor as confidential must be deleted prior to submission.